CLINICAL TRIAL: NCT04649398
Title: Determination of Cerebral Nimodipine Concentrations Following Oral, Intra-venous and Intra-arterial Administration - a Descriptive Pharmacokinetic/Pharmacodynamics Study
Brief Title: Cerebral Nimodipine Concentrations Following Oral, Intra-venous and Intra-arterial Administration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Vienna (Other); Austrian Science Fund (FWF) (Other)
Responsible Party: Principal Investigator, Arthur Hosmann, Principal Investigator, Medical University of Vienna
Other Study IDs: Brain_MD_Nimodipine
Record Dates: First submitted 2020-11-16; First posted 2020-12-02 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Delayed Cerebral Ischemia; Vasospasm, Cerebral
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — Nimodipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, cerebrospinal fluid, microdialysate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- oral nimodipine: 60mg of nimodipine is orally administered every 4 h,
  Interventions: Drug: Nimodipine
- intra-venous nimodipine: nimodipine is continuously administered intra-venously, starting with 0.5 mg/h on day 1 and increased every day for 0.5 mg/h to a maximum dose of 2.0mg/h on day 4
  Interventions: Drug: Nimodipine
- intra-arterial nimodipine: during endovascular procedure 2mg of nimodipine is infused via a microcatheter into the internal carotid artery for 20 minutes
  Interventions: Drug: Nimodipine

INTERVENTIONS:
Drug: Nimodipine — If application of nimodipine is clinically indicated patients will be enrolled in the study protocol according to the inclusion and exclusion criteria. The clinically appropriate route of administration will be administered according to the recommended regimen of the study drug; i.e. within the first 10-14 days intra-venous infusion and thereafter oral administration. Intra-arterial infusion will be performed due to severe cerebral vasospasm with impending stroke.

SUMMARY:
Nimodipine reduces the risk of poor outcome and delayed cerebral ischemia in patients suffering aneurysmal subarachnoid haemorrhage (SAH), but its mode of action is unknown. Its beneficial effect is assumed to be due its neuroprotective effects by reducing intracellular calcium and thereby cellular apoptosis, but higher concentrations might induce marked systemic hypotension, thereby inducing cerebral ischemia. Since several dosing regimes and routes of administration with inconclusive superiority exist and since the target site concentration of nimodipine - the unbound drug concentrations beyond the blood-brain barrier - is still not known, it is reasonable to measure nimodipine concentrations within the blood, cerebrospinal fluid (CSF) and interstitial brain tissue following oral, intra-venous and intra-arterial administration and correlate intra-arterial nimodipine administration to measures of cerebral metabolism and oxygenation.

Therefore, the investigators propose to investigate in 30 patients suffering severe aneurysmal SAH and requiring cerebral microdialysis for cerebral neurochemical monitoring:

* the ability of nimodipine to penetrate into the brain of neurointensive care patients by comparing exposure in brain, CSF and plasma, dependent on the route of administration (i.e. oral, intra-venous, and intra-arterial) and dosing intra-venously (0.5 - 2mg/h)
* the impact of orally, intra-venously, and intra-arterially delivered nimodipine on cerebral metabolism, i.e. lactate/pyruvate ratio, pbtO2 and transcranial doppler flow velocities
* the effect of oral and intra-venous nimodipine on systemic hemodynamic and cardiac parameters, using continuous Pulse Contour Cardiac Output (PiCCO) monitoring
* the penetration properties of ethanol - as an excipient of nimodipine infusion - into the brain by comparing exposure in brain, CSF and plasma and quantifying the neuronal exposure to alcohol dependent on blood levels

ELIGIBILITY:
Inclusion Criteria:

* patient age > 18 years
* aneurysmal subarachnoid hemorrhage
* sedated and mechanically ventilated
* application of brain microdialysis as standard care (due to the severity of subarachnoid haemorrhage or secondary deterioration)
* oral, intra-venous or intra-arterial administration of nimodipine due to clinical indication

Exclusion Criteria:

* contraindication for nimodipine
* no need of intensive care and bedside cerebral microdialysis as standard care
* any disease considered relevant for proper performance of the study or risks to the patient, at the discretion of the investigator

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring intensive care and bedside cerebral microdialysis for cerebral neurochemical monitoring as standard care with a clinical indication for concomitant treatment with either oral, intra-venous or intra-arterial nimodipin
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
cerebral nimodipine concentrations | during the intervention
  Area under the concentration-time curve in brain, cerebrospinal fluid and serum, dependent on the route of administration (i.e. oral, intra-venous, and intra-arterial)
cerebral ethanol concentrations | during the intervention
  Area under the concentration-time curve and maximum concentrations in brain tissue, CSF and blood after intravenous administration

SECONDARY OUTCOMES:
cerebral lactate/pyruvate ratio (LPR) | during the intervention for oral and intravenous administered nimodipine, 12 hours after the intervention for intra-arterial nimodipine administration
  determined by cerebral microdialysis
brain tissue oxygen tension (pbtO2) | during the intervention for oral and intravenous administered nimodipine, 12 hours after the intervention for intra-arterial nimodipine administration
  determined by cerebral parenchymal probes
cardiac output | during the intervention
  measured by Pulse Contour Cardiac Output (PiCCO) monitoring
fluid responsiveness | during the intervention
  measured by Pulse Contour Cardiac Output (PiCCO) monitoring
extravascular lung water index | during the intervention
  measured by Pulse Contour Cardiac Output (PiCCO) monitoring
systemic vascular resistance index | during the intervention
  measured by Pulse Contour Cardiac Output (PiCCO) monitoring
transcranial doppler flow velocities | during the intervention for oral and intravenous administered nimodipine, 12 hours after the intervention for intra-arterial nimodipine administration
  measured in the middle cerebral artery ipsilateral to the microdialysis probe
angiographic vasospasm | immediately after the intervention
  mild: vessel diameter from 60-99%, moderate: vessel diameter from 30-59%, severe: vessel diameter <30% of the physiological lumen
cerebral perfusion pressure | during the intervention for oral and intravenous administered nimodipine, 12 hours after the intervention for intra-arterial nimodipine administration
  measured continuously via intra-arterial and intracranial probes
incidence of delayed ischemic strokes | 3-21 days following subarachnoid haemorrhage
  ischemic strokes on CT scans

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria